CLINICAL TRIAL: NCT04823611
Title: A Phase 1 and 2 Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of AZD8233 Following a Multiple Subcutaneous Dose Administration in Japanese Participants With Dyslipidemia
Brief Title: A Study of AZD8233 in Participants With Dyslipidemia.
Acronym: HAYATE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7990C00006
Record Dates: First submitted 2021-02-01; First posted 2021-04-01 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Dyslipidemia
Keywords: AZD8233; Efficacy; PK; PD; Immunogenicity; Safety; Tolerability
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part A: Single blind Part B: Double blind Part C: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Part A:Placebo (Placebo Comparator): Placebo solution for subcutaneous injection.
  Interventions: Drug: Part A:Placebo
- Part A:AZD8233 (Experimental): AZD8233 for subcutaneous injection.
  Interventions: Drug: Part A:AZD8233
- Part B:Placebo (Placebo Comparator): Placebo solution for subcutaneous injection.
  Interventions: Drug: Part B:Placebo
- Part B:AZD8233 medium dose (Experimental): AZD8233 medium dose for subcutaneous injection.
  Interventions: Drug: Part B:AZD8233
- Part B:AZD8233 low dose (Experimental): AZD8233 low dose for subcutaneous injection.
  Interventions: Drug: Part B:AZD8233
- Part C: Placebo (Placebo Comparator): Placebo solution for subcutaneous injection.
  Interventions: Drug: Part C: Placebo
- Part C: AZD8233 medium dose (Experimental): AZD8233 medium dose for subcutaneous injection.
  Interventions: Drug: Part C: AZD8233

INTERVENTIONS:
Drug: Part A:Placebo — Placebo solution
  Arms: Part A:Placebo
Drug: Part A:AZD8233 — PCSK9-targeted ASO for the reduction of circulating levels of LDL-C.
  Arms: Part A:AZD8233
Drug: Part B:Placebo — Placebo solution
  Arms: Part B:Placebo
Drug: Part B:AZD8233 — PCSK9-targeted ASO for the reduction of circulating levels of LDL-C.
  Arms: Part B:AZD8233 low dose; Part B:AZD8233 medium dose
Drug: Part C: Placebo — Placebo solution
  Arms: Part C: Placebo
Drug: Part C: AZD8233 — PCSK9-targeted ASO for the reduction of circulating levels of LDL-C.
  Arms: Part C: AZD8233 medium dose

SUMMARY:
A Phase 1 and 2 Study of AZD8233 in Participants with Dyslipidemia and this study consists of Part A , Part B and Part C. Part A is designed as a randomized, single-blind (blinding of participants and sites), placebo-controlled, multiple dose, phase 1 study. Part B is designed as a randomized, double-blind, placebo-controlled, dose-ranging, phase 2 study. Part C is designed as a randomized , single-blind (blinding of participants and sites), placebo-controlled, multiple dose, phase 1 study.

DETAILED DESCRIPTION:
Part A: This is designed as a randomized, single-blind (blinding of participants and sites), placebo-controlled, multiple dose, phase 1 study.

Approximately 11 Japanese participants will be randomized in an 8:3 ratio into 1 of the 2 single-blinded treatment arms; AZD8233 high dose or placebo. Participants will be dosed SC on Days 1, 8, 29, and 57.

Part B:This is designed as a randomized, double-blind, placebo-controlled, dose-ranging, phase 2 study. Approximately 60 Japanese participants will be randomized in a 1:1:1 ratio into 1 of the 4 double-blinded treatment arms; AZD8233 low dose, AZD8233 medium dose, or placebo. Participants will be dosed SC on Days 1, 29, and 57.

Part C:This is designed as a randomized, single-blind (blinding of participants and sites), placebo-controlled, multiple dose, phase 1 study.

Approximately 11 Japanese participants will be randomized in an 8:3 ratio into 1 of the 2 single-blinded treatment arms; AZD8233 medium dose or placebo. Participants will be dosed SC on Days 1, 29, and 57.

ELIGIBILITY:
Key Inclusion Criteria:

Part A

* Participants must be 20 to 60 years of age inclusive, at the time of signing the informed consent
* Participants who have a fasting LDL-C ≥ 70 mg/dL but < 140 mg/dL at screening
* Participants who have fasting triglycerides < 400 mg/dL at screening
* Participants who should be receiving statin therapy
* Participants who should be on stable medication for a certain time period prior to randomization
* Body mass index (BMI) between 19 and 40 kg/m2
* Females must not be pregnant and must have a negative pregnancy test at screening and randomisation, must not be lactating , and must be of nonchild-bearing potential

Part B

* Participants must be 20 to 75 years of age inclusive, at the time of signing the informed consent
* Have a fasting LDL-C ≥ 70 mg/dL but < 190 mg/dL at screening (Visit 2)
* Have fasting triglycerides < 400 mg/dL at screening (Visit 2)
* Should be receiving statin therapy
* LDL-lowering medications should be on stable dosing for ≥ 3 months prior to screening with no planned medication or dose change during study participation
* BMI between 19 and 40 kg/m2
* Female participants must not be pregnant and must have a negative pregnancy test at screening and randomisation, must not be lactating, and must not be of childbearing potential

Part C

* Participants must be 20 to 60 years of age inclusive, at the time of signing the informed consent
* Participants who have a fasting LDL-C ≥ 70 mg/dL but < 140 mg/dL at screening
* Participants who have fasting triglycerides < 400 mg/dL at screening
* Participants who should be receiving statin therapy
* Participants who should be on stable medication for a certain time period prior to randomization
* Body mass index (BMI) between 19 and 40 kg/m2
* Females must not be pregnant and must have a negative pregnancy test at screening and randomisation, must not be lactating , and must be of nonchild-bearing potential

Key Exclusion Criteria:

Part A

* eGFR < 60 mL/min/1.73m2 using the Japanese equation
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding. Or participants receiving anti-coagulation therapy
* History of major bleed or high-risk of bleeding diathesis
* Subjects with a high 10-year risk of coronary heart disease as calculated using the Suita score
* Heart rate after 10 minutes of sitting rest < 50 or > 100 beats per minute
* Uncontrolled hypertension defined as sitting SBP > 140 mmHg or DBP > 90 mmHg

Part B

* eGFR < 40 mL/min/1.73m2 using the Japanese equation at Visit 1
* Poorly controlled type 2 diabetes mellitus (T2DM), defined as Haemoglobin A1c (HbA1c) > 10% at Visit 1
* Acute ischaemic cardiovascular event in the last 12 months prior to randomization
* Heart failure with New York Heart Association (NYHA) Class III-IV
* High-risk of bleeding diathesis as judged by the Investigator
* Uncontrolled hypertension defined as sitting SBP > 160 mmHg or DBP > 90 mmHg at Visit 1 or Visit 3
* Heart rate after 10 minutes sitting rest < 50 bpm or > 100 bpm at Visit 1 or Visit 3

Part C

* eGFR < 60 mL/min/1.73m2 using the Japanese equation
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding. Or participants receiving anti-coagulation therapy
* History of major bleed or high-risk of bleeding diathesis
* Subjects with a high 10-year risk of coronary heart disease as calculated using the Suita score
* Heart rate after 10 minutes of sitting rest < 50 or > 100 beats per minute
* Uncontrolled hypertension defined as sitting SBP > 140 mmHg or DBP > 90 mmHg

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Research Site, Chiyoda-ku
  - Research Site, Chūōku
  - Research Site, Osaka
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clewe O, Rekic D, Quartino AL, Carlsson B, Higashimori M, Wernevik L, Hofherr A, Ryden-Bergsten T, Nilsson C, Knochel J. Population pharmacokinetics of a novel PCSK9 antisense oligonucleotide. Br J Clin Pharmacol. 2024 Jun;90(6):1503-1513. doi: 10.1111/bcp.16046. Epub 2024 Mar 19. PMID 38504437
- See also: CSRsynopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00006&attachmentIdentifier=5acc6b71-a65b-42b0-a2b9-9fe64aa7f1c9&fileName=d7990c00006-clinical-study-report-Combined_Redacted.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00006&attachmentIdentifier=eb305a4d-106e-464b-92d0-e179003c58ae&fileName=d7990c00006-sap-part-Combined_redacted_2.pdf&versionIdentifier=
- See also: CSPredacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00006&attachmentIdentifier=225151c3-a0fb-4f5b-8da4-d34867e59881&fileName=d7990c00006-csp-v5_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A:AZD8233 90mg: AZD8233 for subcutaneous injection.
- Part B:AZD8233 50mg; Part C: AZD8233 60mg: AZD8233 medium dose for subcutaneous injection.
- Part B:AZD8233 15mg: AZD8233 low dose for subcutaneous injection.
Period: Overall Study
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Started | 8 | 3 | 22 | 22 | 21 | 8 | 3
Completed (Completed treatment) | 6 | 3 | 21 | 22 | 21 | 8 | 3
Not Completed | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo | Total
Number analyzed (Participants) | 8 | 3 | 22 | 22 | 21 | 8 | 3 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (5.38) | 47.0 (11.36) | 60.6 (6.29) | 64.4 (5.50) | 61.9 (7.04) | 52.0 (6.37) | 52.0 (3.61) | 59.6 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 12 | 7 | 9 | 2 | 0 | 33
  Male | 6 | 2 | 10 | 15 | 12 | 6 | 3 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 8 | 3 | 22 | 22 | 21 | 8 | 3 | 87

OUTCOME MEASURES:

1. Primary Outcome: Part B: Change in LDL-C in Serum at Week 12
Description: Part B: Change from baseline in LDL-C at week 12. Results are based on Mixed Model Repeated Measures (MMRM) analysis on the log-transformed change from baseline. Log-transformed change from baseline is calculated as the visit value in log minus the baseline value in log. The results from the model are then back transformed. Note: log(week 12 data) - log(baseline data) = log(week12/baseline), which is a ratio
Time Frame: Baseline to week 12
Population: Full Analysis Set (Part B only). These data were not pre-specified for parts A and C
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 0 | 0 | 20 | 22 | 21 | 0 | 0
Ratio |  |  | 0.198 [0.167 to 0.235] | 0.458 [0.388 to 0.541] | 0.953 [0.806 to 1.128] |  |

2. Secondary Outcome: Part B: Percentage Change From Baseline in LDL-C in Serum at Week 12
Description: Percentage change from baseline to week 12 in Low-density Lipoprotein Cholesterol (LDL-C) in serum
Time Frame: Measurement at baseline and week 12
Population: Full Analysis Set (Part B only). These data were not pre-specified for parts A and C
Measure: Least Squares Mean (95% Confidence Interval); unit: % change from baseline
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 0 | 0 | 21 | 22 | 21 | 0 | 0
% change from baseline |  |  | -77.13 [-83.67 to -70.59] | -52.48 [-58.85 to -46.11] | -3.24 [-9.68 to 3.19] |  |

3. Secondary Outcome: Part B: Change in PCSK9 in Plasma at Week 12
Description: Part B: Change from baseline in PCSK9 in plasma at week 12. Results are based on Mixed Model Repeated Measures (MMRM) analysis on the log-transformed change from baseline. Log-transformed change from baseline is calculated as the visit value in log minus the baseline value in log. The results from the model are then back transformed. Note: log(week 12 data) - log(baseline data) = log(week12/baseline), which is a ratio
Time Frame: Baseline to week 12
Population: Full Analysis Set (Part B only). These data were not pre-specified for parts A and C
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 0 | 0 | 21 | 22 | 21 | 0 | 0
Ratio |  |  | 0.066 [0.055 to 0.079] | 0.296 [0.248 to 0.352] | 0.874 [0.731 to 1.045] |  |

4. Secondary Outcome: Part B: Percentage Change From Baseline in PCSK9 in Plasma at Week 12
Description: Percentage change from baseline to week 12 in proprotein convertase subtilisin/kexin type-9 (PCSK9) in plasma
Time Frame: Measurement at baseline and week 12
Population: Full Analysis Set (Part B only). These data were not pre-specified for parts A and C
Measure: Least Squares Mean (95% Confidence Interval); unit: % change from baseline
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 0 | 0 | 21 | 22 | 21 | 0 | 0
% change from baseline |  |  | -92.91 [-99.00 to -86.82] | -65.07 [-71.03 to -59.12] | -11.92 [-18.01 to -5.82] |  |

5. Secondary Outcome: Part A & Part C: AUC (0-24) of AZD8233
Description: Area Under the plasma concentration time curve from time 0 to time 24 hours
Time Frame: Day 1 and Day 57
Population: Pharmacokinetic Analysis Set (Parts A and C only). These data were not pre-specified for part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 8 | 0
h.ng/mL
  Day 1 | 5736 (53.55) |  |  |  |  | 3906 (26.56) |
  Day 57 | 5377 (50.57) |  |  |  |  | 3493 (32.47) |

6. Secondary Outcome: Part A & Part C: Cmax of AZD8233
Description: Maximum plasma concentration
Time Frame: Day 1 and Day 57
Population: Pharmacokinetic Analysis Set (Parts A and C only). These data were not pre-specified for part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 8 | 0
ng/mL
  Day 1 | 1525 (62.11) |  |  |  |  | 830.8 (23.90) |
  Day 57 | 1271 (70.63) |  |  |  |  | 781.2 (50.34) |

7. Secondary Outcome: Part A & Part C: t1/2 of AZD8233
Description: Terminal half-life
Time Frame: Day 1 and Day 57
Population: Pharmacokinetic Analysis Set (Parts A and C only). These data were not pre-specified for part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 8 | 0
hours
  Day 1 | 3.459 (45.69) |  |  |  |  | 2.751 (35.94) |
  Day 57 | 2.848 (44.73) |  |  |  |  | 2.527 (28.36) |

8. Secondary Outcome: Part A & Part C: CL/F (L/h) of AZD8233
Description: Apparent plasma clearance
Time Frame: Day 1 and Day 57
Population: Pharmacokinetic Analysis Set (Parts A and C only). These data were not pre-specified for part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 8 | 0
L/h
  Day 1 | 15.58 (52.84) |  |  |  |  | 15.31 (26.36) |
  Day 57 | 16.62 (50.44) |  |  |  |  | 17.14 (32.25) |

9. Secondary Outcome: Part A & Part C: Vz/F (L)
Description: Apparent Volume of distribution during the terminal phase
Time Frame: Day 1 and Day 57
Population: Pharmacokinetic Analysis Set (Parts A and C only). These data were not pre-specified for part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 8 | 0
L
  Day 1 | 77.74 (106.7) |  |  |  |  | 60.77 (56.66) |
  Day 57 | 68.30 (58.04) |  |  |  |  | 62.49 (56.80) |

ADVERSE EVENTS:
Time Frame: From date of first dose, throughout treatment period and including follow-up period, 24 weeks for Parts A, B and C.
Description: MedDRA 24.1 for Part A, MedDRA 25.0 for Parts B & C
Arm/Group | Part A:AZD8233 90mg | Part A:Placebo | Part B:AZD8233 50mg | Part B:AZD8233 15mg | Part B:Placebo | Part C: AZD8233 60mg | Part C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/22 | 0/22 | 0/21 | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/22 | 0/22 | 0/21 | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 6/8 | 2/3 | 5/22 | 6/22 | 7/21 | 2/8 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A:AZD8233 90mg (N=8) | Part A:Placebo (N=3) | Part B:AZD8233 50mg (N=22) | Part B:AZD8233 15mg (N=22) | Part B:Placebo (N=21) | Part C: AZD8233 60mg (N=8) | Part C: Placebo (N=3)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT04823611/Prot_008.pdf
  • Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT04823611/SAP_009.pdf